CLINICAL TRIAL: NCT04719468
Title: Efficacy of Ballet Dancing on Motor and Non-motor Symptoms of Parkinson's Disease: a Hybrid Type 2 Effectiveness-implementation Trial
Brief Title: PD-Ballet: Effectiveness and Implementation in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 275588
Record Dates: First submitted 2020-07-23; First posted 2021-01-22 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
Keywords: dance; ballet; complementary therapy; exercise; multimodal
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded rater
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Dance with ballet elements
- Usual Treatment (No Intervention): usual treatment with the addition of joining 'Tea and Biscuit' sessions remotely

INTERVENTIONS:
Other: Dance with ballet elements — Ballet-based dance sessions will be delivered by trained artists within the English National Ballet group in a professional dance space/ delivered remotely, COVID-19 permitting.
  Arms: Intervention

SUMMARY:
Current literature consistently demonstrates beneficial motor effects of dance-based therapies in Parkinson's disease, along with improved quality of life. Little is known about the non-motor gains following such therapy. To date, no RTC has been conducted to investigate the benefits of ballet dancing in Parkinson's disease.

The investigators aim to recruit 160 people with Parkinson's to either: participate in a 12-week ballet-based dancing intervention followed by a 'social Tea and Biscuit' session, or 12-week usual treatment monitoring and 'social Tea and Biscuit' sessions taking place after each intervention session. This study employs a randomised, controlled, single-blind, hybrid type 2 design with a hybrid implementation protocol to investigate both clinical efficacy of the programme and implementation aspects. The project's primary outcome measure is centered around non-motor symptoms of PD. Other measures include motor assessments, wearable sensors and quality of life assessments.

Due to COVID-19 pandemic, the delivery of the sessions will be a hybrid model - virtual sessions will be the primary method, with some capacity for in-person delivery when possible and deemed safe.

DETAILED DESCRIPTION:
Parkinson's Disease is a neurodegenerative condition currently affecting over 120,000 people in the UK and this number is set to double by 2065. The current treatment is based around symptomatic pharmacotherapy with levodopa being the gold standard. Currently there is some evidence for non-pharmacological treatments outlined by NICE guidelines, with no recommendations to specific adjuvant non-pharmacotherapies to aid PD symptoms, other than referral for physiotherapy. However, physical exercise has been shown to improve balance, strength, coordination and gait, leading to a significant improvement in quality of life.

While a clear benefit of physical exercise on the motor symptoms is evident, few studies to date focused on the effects of group classes and on non-motor effects. Dance is emerging as a therapeutic option with cognitive, functional and psychosocial benefits, due to it being a multi-dimensional activity offering auditory, visual and sensory stimulation, musical experience, social interaction, memory, motor learning and emotional perception, expression and interaction and as such stimulating multiple pathways. To date, no research has explored acute and chronic effects of exercise based interventions (such as dance therapy with ballet) in comparison to the conventional therapy-based management of Parkinson's.

This is a randomised, controlled, single-blind study involving 160 PwP across all stages of the disease. Participants will be allocated to either standard therapy plus 12 weekly sessions of ballet-based dancing followed by 'Tea and Biscuit' session or standard therapy with 'Tea and Biscuit' session on a 2:1 ratio. Non-motor symptoms, motor symptoms and quality of life will be measured using validated scales, questionnaires and wearable sensor recordings (Parkinson's KinetiGraph, GaitSmart). Furthermore, electrophysiological measures will be performed to determine the effects on cortical activity in a subgroup of participants. Assessments will be performed by a blinded rater at baseline and at the end of the intervention. The project will also explore the possibility of implementation of such therapy into the current pathways.

Due to COVID-19 pandemic, the delivery of the sessions will be a hybrid model - virtual sessions will be the primary method, with some capacity for in-person delivery when possible and deemed safe.

ELIGIBILITY:
Effectiveness investigation eligibility criteria (PwPs only)

1. Inclusion:

   * Age of 18 and upwards
   * diagnosis of idiopathic Parkinson's disease (PD) according to the UK PD Brain Bank criteria
   * Hoehn Yarhr stages I-V
2. Exclusion:

   * diagnosis or suspicion of other causes for parkinsonism
   * advanced-stage therapy consideration (deep brain stimulation, continuous levodopa duodenal infusion, and continuous subcutaneous apomorphine infusion)
   * any condition interfering with the ability to give the informed consent
   * Indication of dementia through a score of ≤21 on MoCA
   * enrolment in a simultaneous investigational trial
   * inability to travel to the weekly sessions

Implementation science investigation eligibility criteria f) Inclusion:

* People with Parkinson's - patients with a formal diagnosis of PD who have participated in the PD-Ballet intervention.
* Family members of PwP - relatives/carers/nominated person of the patients with a formal diagnosis of PD who have participated in the PD-Ballet intervention
* Clinicians (Referrers) - neurologists/geriatricians/neuropsychiatrists/SALT/OT, as well as PD specialist nurses, physicians and research staff experienced in PD
* Dance leaders (Deliverers) - English National Ballet dancers involved in the PD-Ballet project
* Support staff (Supporters)- other parties involved with the PD-Ballet project

  g) Exclusion:
* People with Parkinson's - parkinsonism other than PD, lack of involvement in the PD-Ballet project
* Clinicians - Neurologists/geriatricians/neuropsychiatrists/SALT/OT, as well as PD specialist nurses, physicians and research staff experienced in PD
* Dance leaders - English National Ballet dancers not involved in the PD-Ballet project
* Support staff - other parties not involved with the PD-Ballet project

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in total score of the Movement Disorders Society Sponsored Non-Motor Rating Scale | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness Primary Outcome Measure, higher score indicate worse non-motor symptomatology, the maximum score is 1008.
Acceptability of Intervention Measure | post intervention (week 12)
  Implementation Effectiveness Primary Outcome Measure - a 4 item, 5-point likert scale

SECONDARY OUTCOMES:
Change in total score of the Unified Parkinson's Disease Rating Scale | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A higher score indicates worse motor condition
Change in total score of 10-meter walk test | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. Time taken to walk 10 meters is calculated and compared at specific timepoints.
Change in total score of King's Parkinson's Pain Scale | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A higher score indicates worse levels of pain
Change in total score of Timed Up and Go test | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. Time taken to carry out the test measured. A change between timepoints will be measured.
Change in total score of Montreal Cognitive Assessment | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. Maximum score 30. Lower scores indicate cognitive impairment.
Clinical Impression of Severity Index for Parkinson's disease | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  provides a clinical judgment on Parkinson's disease (PD) severity based on motor symptoms and complications, cognitive status, and disability
Change in total score of Parkinson's Disease Sleep Scale 2 | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. Higher score indicates worse sleep quality
Change in total score of Parkinson's Disease Questionnaire-8 | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A higher score indicates worse quality of life.
Change in total score and sub-scores of Hospital Anxiety and Depression Scale | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. Higher score indicates worse anxiety and depression.
Change in total score of Schwab and England Scale | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A higher score indicates higher level of independence in performing activities of daily living.
Change in total score of EQ-5D-5L questionnaire | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A lower score indicates better quality of life
Change in total score of Parkinson's Fatigue Scale-16 | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A higher score indicates more fatigue.
Change in total score of Physical Activity Scale for the Elderly | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A higher score indicates more activity
Change in total score of Starkstein Apathy Scale | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. Higher score indicates more apathy.
Change in total score of Wearing Off Questionnaire-9 | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. Higher score indicates worse wearing-off.
Change in total score of Zaritt Burden Interview | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness. A higher score indicates more carer burden.
Electrodiagnostic Measures - Transcranial Magnetic Stimulation paired with Electroencephalography and electromyography. | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness - exploratory measure. EMG data are analysed via Spike2 software (Cambridge Electronic Design). Peak-to-peak MEP amplitudes are measured for each trial and averaged per condition. SICI is calculated as the ratio of mean conditioned MEP to mean unconditioned MEP. TMS-evoked EEG potentials will be calculated by averaging artifact-free EEG trials for each experimental condition (i.e., before and after intervention). To smooth the signal a low-pass filter of 45 Hz will be applied to TEPs. The aim is to evaluate drug-induced changes for the 5 typical TEPs components (P = Positive, N = Negative) in accordance with the literature: N15-P25, N45, P70, N100, and P180.
Change in the scores of Parkinson's KinetiGraph parameters (bradykinesia, dyskinesia, tremor, immobility) | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Clinical Effectiveness, objective artigraphy based wearable sensor worn at home for 6 days at each time point.
Feasibility of Intervention Measure (FIM) | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Implementation Effectiveness - a 4-item, 5-point likert scale
Intervention Appropriateness Measure (IAM) | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Implementation Effectiveness - a 4-item, 5-point likert scale
Sustainability scale (NOMAD) | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Implementation Effectiveness - a 19 item implementation science survey (Finch et al., 2015)
Implementation costs | Baseline (week -4 to 0), end of intervention (week 12-14) and up to 24 weeks post intervention depending on participant availability
  Health Economics - questionnaire regarding the potentially incurred costs related to clinical care for a person with Parkinson. The investigators will measure the potential change in direct and indirect costs incurred from clinical care.

CONTACTS AND LOCATIONS:
Overall Officials: K Ray Chaudhuri, Professor, Principal Investigator — King's College London
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Podlewska AM, Batzu L, Soukup T, Sevdalis N, Bakolis I, Derbyshire-Fox F, Hartley A, Healey A, Woods A, Crane N, Pariante C, Ray Chaudhuri K. The PD-Ballet study: study protocol for a randomised controlled single-blind hybrid type 2 clinical trial evaluating the effects of ballet dancing on motor and non-motor symptoms in Parkinson's disease. BMC Complement Med Ther. 2024 Jan 17;24(1):41. doi: 10.1186/s12906-023-04296-y. PMID 38233784
- [Derived] Soukup T, Davis RE, Baldellou Lopez M, Healey A, Estevao C, Fancourt D, Dazzan P, Pariante C, Dye H, Osborn T, Bind R, Sawyer K, Rebecchini L, Hazelgrove K, Burton A, Manoharan M, Perkins R, Podlewska A, Chaudhuri R, Derbyshire-Fox F, Hartley A, Woods A, Crane N, Bakolis I, Sevdalis N. Study protocol: randomised controlled hybrid type 2 trial evaluating the scale-up of two arts interventions for postnatal depression and Parkinson's disease. BMJ Open. 2022 Feb 1;12(2):e055691. doi: 10.1136/bmjopen-2021-055691. PMID 35105591